CLINICAL TRIAL: NCT03807180
Title: Tai Chi in Patients With Ankylosing Spondylitis
Brief Title: Effects of Tai Chi in Patients With Ankylosing Spondylitis Receiving Anti-tumor Necrosis Factor Alpha Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Bilge Basakci Calik, Assoc Prof, PT, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 60116787-020/55441
Record Dates: First submitted 2019-01-10; First posted 2019-01-16 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Spondylitis, Ankylosing
Keywords: Tai Chi; ankylosing spondylitis; functionality
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Tai Ji; Exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled
Who Masked: Participant
Masking Description: Patients with Ankylosing spondylitis receiving anti-tnf alpha therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of Tai Chi (Other): Group of Tai Chi intervention include 18 patients with AS. Tai Chi exercise method, which is composed of combination of physical exercise and relaxation techniques, will be applied by an experienced physiotherapist who is trained with Tai Chi. The training will take 60 minutes, 2 days a week and 10 weeks in total.
  Interventions: Other: Tai Chi (exercise)
- Group of control (No Intervention): Conventional exercises are stretching for the cervical, thoracic and lumbar flexibility, shoulder circumference, hamstring and erector spinal muscles, strengthening exercises for abdominal, back and proximal muscles. The exercises that will be taught in detail to each stage of the patient will be performed at home by the patient for 60 minutes, 2 days a week. The patients will be inspected and controlled by monthly controls.

INTERVENTIONS:
Other: Tai Chi (exercise) — Tai Chi exercise method, which is composed of combination of physical exercise and relaxation techniques for patients with rheumatic diseases.
  Arms: Group of Tai Chi

SUMMARY:
Ankylosing Spondylitis (AS) is a chronic inflammatory rheumatic disease that causes a decrease in physical activity, fatigue, sleep problems and psychological consequences such as depression, anxiety and stress by primarily affecting the sacroiliac joint and spine. The aim of the treatment of AS is to prevent the hardness and flexion deformity associated with the disease; to maintain the patient's healthy psychological and physical condition. The first step in the treatment of AS; Pharmacological treatment of NSAIDs or Anti-TNFs along with exercise. Exercise, especially pain and immobility symptoms control provides patients with disease is an advantage.

Tai Chi Chuan or Taiji is a traditional Chinese exercise method that has been applied for more than 300 years. Exercises based on Chinese medicine and martial arts. It is a combination of physical exercise and relaxation techniques and is used to improve the mental and physical health of individuals. In literature, balance, strength, coordination, postural control, agility, reaction time, flexibility has attracted attention for developing such factors. In addition, it increases muscle strength in elderly people and decreases the risk of falling; Rheumatoid arthritis and Osteoarthritis-related symptoms have been reported to improve in a positive way. In the literature, there is only one study examining the efficacy of Tai Chi in AS patients. According to the results of this study, Tai Chi has a positive effect on disease activity and flexibility of patients with AS.

Although there is consensus on exercise role in the treatment of AS, when the literature is reviewed, it is seen that the strict and definite guidelines on the type and frequency of exercises are not yet described. There is no defined protocol for which specific exercise is appropriate in AS. The literature considers that more information is needed on the various physical therapy programs related to intensity, frequency and duration to determine the most appropriate activity for the disease.

The aim of this study was to investigate the effect of Tai Chi exercises on functionality, disease activity, functional exercise capacity, spinal mobility, lower extremity strength and quality of life in AS patients with biological agents.

DETAILED DESCRIPTION:
At least 36 AS patients followed-up by Antalya Training and Research Hospital, who are receiving Anti-TNF therapy and who do not have any other disease affecting their functions will be included in the study. There were 18 patients in the conventional treatment group and 18 patients in the Tai Chi group.

After the demographic data of AS patients were recorded, Bath AS Disease Activity Index (BASDAI), Bath AS Disease Activity Index (BASFI) and Bath AS Metrology Index (BASMI), respectively, to be used for activity and basic measurements of the disease, 6 minutes walking test to measure aerobic capacity , Cognitive Exercise Therapy Approach Scale and Ankylosing Spondylitis Quality of Life Questionnaire to be used for quality of life, 30 second sit-down test to evaluate the lower extremity strength. In addition, 10-20 ml (1-2 tubes) of blood will be taken from the patient's arm, the amount of substances such as erythrocyte sedimentation rate (ESR) and C reactive protein (CRP) in the blood will be measured. Patients will not be charged any fee related to this process. Evaluation methods will be applied to the cases before the start of training and after the completion of the training.

For the training, both patient groups were randomly divided into two groups: the first group was treated with conventional treatment and the second group with Tai Chi training. The training will last 10 weeks.

Conventional treatment; stretching for the cervical, thoracic and lumbar flexibility, shoulder circumference, hamstring and erector spinal muscles, strengthening exercises for abdominal, back and proximal muscles. The exercises that will be taught in detail to each stage of the patient will be performed at home by the patient for 60 minutes, 2 days a week. The patients will be inspected and controlled by monthly controls.

Tai Chi exercise method, which is composed of combination of physical exercise and relaxation techniques, will be applied by an experienced physiotherapist who is trained with Tai Chi. The training will take 60 minutes, 2 days a week and 10 weeks in total.

ELIGIBILITY:
Inclusion Criteria:

* Being sedentary (not routinely involved in exercise activities during the last 3 months).
* We have been using fixed dose medication for at least 6 months (no change in drug treatment during the study).
* No communication problem

Exclusion Criteria:

* Functional disorders more effective than ankylosing spondylitis;
* Diastolic heart failure
* Renal failure
* Severe asthma knee osteoarthritis
* Metastatic prostate cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Bath Ankylosing Spondylitis Functional Index (BASFI) | ten weeks
  This self-assessment instrument was designed by a team of medical professionals in conjunction with patients, and consists of 8 specific questions regarding function in AS and 2 questions reflecting the patient's ability to cope with everyday life. Each question is answered on a 10 cm horizontal visual analog scale, the mean of which gives the BASFI score (0-10). Higher scores show poor functionality.
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | ten weeks
  The index, designed by a multidisciplinary team with input from patients, consists of six 10 cm horizontal visual analog scales to measure severity of fatigue, spinal and peripheral joint pain, localized tenderness and morning stiffness (both qualitative and quantitative). The final BASDAI score has a range of 0 to 10. Higher scores show poor disease activity.
Bath Ankylosing Spondylitis Metrology Index (BASMI) | ten weeks
  İt is for quantify the mobility of the axial skeleton in ankylosing spondylitis (AS) patients and allow objective assessment of clinically significant changes in spinal movement.It is included of clinical measures of cervical rotation, tragus to wall distance, lumbar flexion, lumbar side flexion, and intermalleolar distance.Each item is scored from 0-10 based on individually defined cut points. Ranges are given as cervical rotation (>85.0° to ≤8.5°), tragus to wall (<10 cm to ≥38 cm), lumbar flexion (>7.0 cm to ≤0.7 cm), lumbar side flexion (>20.0 cm to <1.2 cm), and intermalleolar distance (≥120 cm to <30 cm). Higher scores show poor spinal mobility.

SECONDARY OUTCOMES:
Ankylosing Spondylitis Life Quality Questionnaire (ASQol), | ten weeks
  It is purpose to measure the impact of ankylosing spondylitis (AS) on health-related quality of life from the patient's perspective.The questionnaire includes items related to the impact of disease on sleep, mood, motivation, coping, activities of daily living, independence, relationships, and social life. It is included 18 items.Dichotomous responses, with 0 scored for a "no" and 1 scored for a "yes" for each item. Total score is the sum of the individual responses.Score range is 0-18, with higher scores reflecting greater impairment of health-related quality of life.
6 minute walking test | ten week
  The maximum distance that individuals can walk in a 30-meter straight and inclined corridor for 6 minutes is recorded. Higher distances show better aerobic capacity

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Ayan, Dr, Study Chair — Antalya Training and Research Hospital
Locations (1):
- Antalya Education and Research Hospital, Antalya, Konyaalti, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will use Statistical package for the social sciences (SPSS) for participant data after interventions

REFERENCES:
- [Result] Lee EN, Kim YH, Chung WT, Lee MS. Tai chi for disease activity and flexibility in patients with ankylosing spondylitis--a controlled clinical trial. Evid Based Complement Alternat Med. 2008 Dec;5(4):457-62. doi: 10.1093/ecam/nem048. Epub 2007 Jul 13. PMID 18955296